CLINICAL TRIAL: NCT06379269
Title: Effectiveness Verification of a Smartphone-based System for Assessment and Health Care on Myofascial Pain Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Cheng Kung University (Other); National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, Li-Wei Chou, Doctor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH112-REC3-160
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Myofascial Pain Syndrome
Keywords: myofascial pain syndrome; smartphone
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App group (Experimental)
  Interventions: Device: App healthcare
- Control group (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Device: App healthcare — Self-developed app: includes home stretching and strengthening exercises, muscle release technique instruction.
  Arms: App group
Other: Control — general education and home rehab program
  Arms: Control group

SUMMARY:
Myofascial pain syndrome (MPS) is the most common musculoskeletal pain disorder. The pain originates from myofascial trigger points (TrPs) in skeletal muscle. The muscle that presents with TrPs would be identified through clinical diagnosis and assessment, and further treatment would be designed according to the identified muscle.With the high penetration rate of smartphones, it would be convenient to utilize smartphones as the assistive technology in the assessment and intervention of MPS. The smartphone-based MPS assessment and care system could eliminate the restrictions of the epidemic, and provide an independent usage, precisely identifying muscle with TrPs and personalized care plan application. Therefore, the purpose of this study is to 1. develop a smartphone-based assessment and health care system for patients with myofascial pain syndrome. And to 2. verify the feasibility and validity of the system assessment function. And to 3. testify the effectiveness of the system health care functions for patient intervention.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is the most common musculoskeletal pain disorder. The pain originates from myofascial trigger points (TrPs) in skeletal muscle. The muscle that presents with TrPs would be identified through clinical diagnosis and assessment, and further treatment would be designed according to the identified muscle. Common treatments include medications, dry needles, and physical therapy. Among them, physical therapy aims to treat the involved muscle. With the advancement of technology, mHealth (mobile health) has been gradually developed in recent years. With the high penetration rate of smartphones, it would be convenient to utilize smartphones as the assistive technology in the assessment and intervention of MPS. The smartphone-based MPS assessment and care system could eliminate the restrictions of the epidemic, and provide an independent usage, precisely identifying muscle with TrPs and personalized care plan application. Therefore, the purpose of this study is to 1. develop a smartphone-based assessment and health care system for patients with myofascial pain syndrome. And to 2. verify the feasibility and validity of the system assessment function. And to 3. testify the effectiveness of the system health care functions for patient intervention.Methods: Feasibility evaluation: Subjects with MPS will be recruited to perform the assessment of the system on their own. And the assessment results for the system will be compared with clinical assessment results done by a rehabilitation physician. The feasibility of the smartphone app will be analyzed through the system usability scale.Health care effects evaluation: Subjects with MPS will be recruited and randomly assigned to the intervention group and control group. The intervention group will receive the smartphone app health care program, and the control group will receive health education. Outcomes will be measured before and after the intervention. The training effects of the app will be evaluated by comparing it with the control group.Expected Results & Contribution: The smartphone app for identifying the muscle presenting TrPs on MPS subjects is feasible. The healthcare effects of the smartphone app for MPS subjects are effective. Offering an easy-used and effective tool for clinicians and subjects with MPS to evaluate and improve pain and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* For those diagnosed with myofascial pain syndrome by a rehabilitation physician, the diagnostic conditions meet the five major signs, including:

  1. Regional pain,
  2. Transfer pain,
  3. Muscle tight band,
  4. Tender points in the tight band. ,
  5. Limitation of joint mobility,
* And symptoms consistent with any of the items, including:

  1. Complaints of pain that appear after applying pressure on tender points,
  2. Local throbbing reaction,
  3. Pain disappears after injection or after stretching

Exclusion Criteria:

* Have any neurological diseases that may cause pain,
* have a history of surgery in the past six months,
* the affected area is in a state of acute inflammation,
* have open wounds, etc.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
current pain visual analogue scale | 10 minutes
  pain will be evaluated with visual analogue scale(VAS). 0 means no pain at all;10 means extremely painful.

SECONDARY OUTCOMES:
functional questionnaire | 20 minutes
  corresponding functional questionnaire to the specific body part of the subject. For the neck area, the Neck Disability Index is used. The higher the score, the more disability the patient is. For the lower back area, the Oswestry Disability Index is used. The higher the score, the more disability the patient is. For the upper limb, the Disability of the Arm, Shoulder, and Hand is used. The higher the score, the more severe the patient is. For the lower limb, the Lower Extremity Functional Scale is used. The higher the score, the more sever the patient is.